CLINICAL TRIAL: NCT01469338
Title: A Phase II Clinical Trial of Cabazitaxel Plus Prednisone With Octreotide in the Treatment of Castration-Resistant Prostate Cancer (CRPC) Previously Treated With Docetaxel
Brief Title: Cabazitaxel Plus Prednisone With Octreotide For Castration-Resistant Prostate Cancer (CRPC) Previously Treated With Docetaxel
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 4P-11-3; NCI-2011-03266 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-11-01; First posted 2011-11-10 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Diarrhea; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Diarrhea; Prostatic Neoplasms | interventions — cabazitaxel; XRP6258; Prednisone; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (management of therapy complications) (Experimental): Patients receive cabazitaxel IV over 1 hour on day 1, prednisone PO QD, and octreotide pamoate IM on day 1. Patients also receive octreotide acetate SC TID on days 1-14 of course 1 only. Treatment with cabazitaxel repeats every 21 days and treatment with prednisone and octreotide pamoate repeats every 4 weeks for up to 10 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cabazitaxel; Drug: prednisone; Drug: octreotide pamoate; Other: questionnaire administration; Drug: octreotide acetate

INTERVENTIONS:
Drug: cabazitaxel — Given IV
  Other Names: Jevtana; RPR-116258A; taxoid XRP6258; XRP6258
Drug: prednisone — Given PO
  Other Names: DeCortin; Deltra
Drug: octreotide pamoate — Given IM
  Other Names: OP LAR; Sandostatin pamoate; Sandostatin pamoate LAR; SMS 201-995 pa; SMS 201-995 pa LAR
Other: questionnaire administration — Ancillary studies
Drug: octreotide acetate — Given SC
  Other Names: Longastatin; Longastatina; Samilstin; SMS 201-995

SUMMARY:
This phase II trial studies how well octreotide works in reducing diarrhea in patients receiving cabazitaxel and prednisone for hormone-resistant prostate cancer (HRPC) previously treated with docetaxel. Octreotide may prevent diarrhea by blocking the secretion of several hormones in patients receiving chemotherapy for prostate cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the impact of octreotide in reducing the incidence of grade 2 or greater diarrhea in men receiving cabazitaxel plus prednisone for castration-resistant prostate cancer (CRPC) after docetaxel therapy.

SECONDARY OBJECTIVES:

I. Overall survival (OS).

II. Progression-free survival (PFS) (defined as the time between treatment start and the first date of progression as measured by objective tumor progression using the Response Evaluation Criteria In Solid Tumors (RECIST), pain progression or death).

III. Prostate-specific antigen (PSA) response rate.

IV. Objective response rate.

V. Pain response.

VI. Toxicity.

OUTLINE:

Patients receive cabazitaxel as intravenous (IV) infusion over 1 hour on day 1, prednisone by mouth (PO) every day (QD), and octreotide pamoate given as intramuscular (IM) injection on day 1. Patients also receive octreotide acetate as a subcutaneous (SC) injection three times a day (TID) on days 1-14 of course 1 only. Treatment with cabazitaxel repeats every 21 days and treatment with prednisone and octreotide pamoate repeats every 4 weeks for up to 10 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up at 1 month, every 3 months until disease progression, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed prostate cancer
* Measurable disease on computed tomography (CT) or evaluable disease with an elevated PSA
* Documented progression on (a) at least one prior hormone treatment, which must have incorporated luteinizing hormone-releasing hormone (LHRH) agonist therapy AND (b) at least one chemotherapy regimen, which must have included docetaxel; progression may be demonstrated by radiologic criteria or by PSA only if accompanied by new or worsening symptoms (pain progression)
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-2
* Absolute neutrophil count (ANC) more than or equal to 1500/ul
* Hemoglobin more than or equal to 8.0 g/dL
* Platelet count more than or equal to 100,000/ul
* Serum creatinine less than or equal to 1.5x the upper limit of normal (ULN)
* Bilirubin less than or equal to ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 1.5x ULN
* Must be recovered from acute and late effects of any prior surgery, radiotherapy or other anti-neoplastic therapy
* Patients or their legal representatives must be able to read, understand, and provide informed consent
* Men of childbearing potential must consent to use barrier contraception while on treatment and for 90 days thereafter
* Palliative radiation for metastatic disease is allowed if less or equal to 40% of the total bone marrow was irradiated; 28 days must have elapsed since completion of radiation therapy (RT) with bone marrow recovery; soft tissue disease irradiated in the prior 2 months may not be designated as measurable disease
* Concomitant bisphosphonate use is permitted if the dose had been stable for 12 weeks prior to enrollment

Exclusion Criteria:

* Treatment with radiotherapy, chemotherapy or any investigational agent in the prior 4 weeks
* Major surgery in the prior 4 weeks
* Prior treatment with cabazitaxel
* Patients with known hypersensitivity to cabazitaxel, other drugs formulated with polysorbate 80 or octreotide
* Inability to tolerate oral prednisone
* Grade 2 or greater diarrhea in the prior 2 weeks
* Grade 2 or greater neuropathy or stomatitis
* Presence of an active uncontrolled infection or fever greater or equal to 38.5 degrees
* Presence of parenchymal brain metastases; patients with neurological symptoms must have a CT or magnetic resonance imaging (MRI) of the brain showing no metastases within 60 days of enrollment
* Prior malignancy within the past 5 years with the exception of curatively treated basal cell or squamous cell carcinoma of the skin or superficial bladder or other stage I or stage II cancer in complete remission for at least 12 months
* History of unstable or newly diagnosed angina pectoris, documented history of current serious arrhythmia or congestive heart failure (CHF) or recent myocardial infarction (MI)within 6 months of enrollment
* Known human immunodeficiency virus (HIV) or hepatitis infection
* Life expectancy less than 3 months
* Presence of any other medical condition, including mental illness or substance abuse, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with interpretation of the results
* Lack of ability/willingness to give informed consent
* Lack of ability/willingness to receive octreotide injection
* Anticipated non-availability for study visits/procedures
* Patients with uncontrolled diabetes, defined as a HbA1c greater than 7% or greater or equal to 8% despite therapy, or a fasting plasma glucose more than 2x ULN; at the investigator's discretion, non-eligible patients can be re-screened after adequate medical therapy has been instituted

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-07; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Development of Grade 2 plus diarrhea | Baseline through 21 days after the last administration of cabazitaxel
  Defined by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 criteria as an increase in frequency of 4 or greater stools per day over baseline, incontinence, diarrhea warranting hospitalization or diarrhea limiting self-care activities of daily living (ADL). Baseline frequency will be defined in the pre-treatment assessment from cycle 1 as the maximum number of stools in one 24 hour period during the past 2 weeks. Any incidence of grade 2 or greater diarrhea during treatment or for up to 21 days after the last administration of cabazitaxel will be included in this endpoint.

SECONDARY OUTCOMES:
Progression-Free Survival | At 1 month after completion of treatment, every 3 months until disease progression, and then every 6 months thereafter
Overall Survival | At 1 month after completion of treatment, every 3 months until disease progression, and then every 6 months thereafter
RECIST response for patients with measurable disease | Baseline, after every 4 courses, at the end of treatment, and then every 6 months
Prostate-Specific Antigen response | Baseline, day 1 of each course, at the end of treatment, and then every 6 months
Pain palliation in patients with a baseline pain score greater or equal to 2 | Baseline, day 1 of each 3 week course, at the end of treatment, and then every 6 months for up to 52 weeks
Toxicity (adverse events considered to be at least possibly drug-related) | Baseline, day 1 of each course, and at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Pinski, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States